CLINICAL TRIAL: NCT06812364
Title: COMPARISON OF THE EFFICACY OF ONE LEVEL AND TWO LEVEL OF BILATERAL THORACIC ERECTOR SPINAE PLANE BLOCK COMBINED WITH GENERAL ANESTHESIA IN LAPAROSCOPIC BARIATRIC SURGERY FOR OBESE PATIENTS: RANDOMIZED CONTROLLED TRIAL
Brief Title: Bilateral Thorathic Erector Spinae Plane Block in Laparoscopic Bariatic Surgeries
Acronym: ESPBbariatrics
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Belal Galal Mostafa Mohammed Khater, Assistant lecturer, Cairo University
Other Study IDs: MD-407-2024
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain Relief
Keywords: one level ESPB; two level ESPB; bariatric surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- One level ESPB: Ultrasound will be sagittal placed against the target vertebral level T7 vertebrae in the lateral or sitting position and moved in approximately 3-cm lateral to the spinous process. The Erector Spinae muscle and transverse process will be then identified, and a blunted tip ,100mm, 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be advanced, using the in-plane approach, in caudal -to- cephalad direction, through the inter fascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane, and on injection of 3 ml normal saline to confirm the correct needle tip position. The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (30mL into each side) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the T7 vertebrae
  Interventions: Procedure: one level ESPB
- two level ESPB: The target vertebral levels are T5 transverse process (at the level of Sternal Angle, above T7 by tow vertebra) and T10 transverse process (at the level of Xiphisternal Junction, below T7 by 3 vertebrae).
  The block will be performed bilaterally by injecting 60mL of 0.25% bupivacaine (15mL into each of four site) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the thoracic vertebrae 5 and 10 (at the most lateral part of the transverse process) in the same technique
  Interventions: Procedure: two level ESPB

INTERVENTIONS:
Procedure: one level ESPB — Ultrasound will be sagittal placed against the target vertebral level T7 vertebrae in the lateral or sitting position and moved in approximately 3-cm lateral to the spinous process. The Erector Spinae muscle and transverse process will be then identified, and a blunted tip ,100mm, 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be advanced, using the in-plane approach, in caudal -to- cephalad direction, through the inter fascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane, and on injection of 3 ml normal saline to confirm the correct needle tip position. The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (30mL into each side) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the T7 vertebrae
  Groups: One level ESPB
Procedure: two level ESPB — The target vertebral levels are T5 transverse process (at the level of Sternal Angle, above T7 by tow vertebra)(19) and T10 transverse process (at the level of Xiphisternal Junction, below T7 by 3 vertebrae).
  The block will be performed bilaterally by injecting 60mL of 0.25% bupivacaine (15mL into each of four site) into the fascial plane between the deep surface of the Erector Spinae muscle and the bilateral transverse processes of the thoracic vertebrae 5 and 10 (at the most lateral part of the transverse process) in the same technique.
  Groups: two level ESPB

SUMMARY:
The study is to evaluate effectiveness of one-level versus two-level thoracic ESP block on intraoperative and postoperative analgesia in bariatric surgeries and to compare total opioid consumption of both groups.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity is steadily increasing. The epidemic of overweight and obesity presents a major challenge to chronic disease prevention and health across the life course around the world.

Bariatric surgery has proved to be an efficient intervention in the management of obesity. As a result, the number of post-bariatric surgery patients in the population is growing .

Postoperative pain is categorized into acute pain which occur immediately after surgery (up to 7 days) and chronic pain which lasts more than 3 months after the injury . Laparoscopic bariatric surgery often presents significant pain, ranging from moderate to severe, particularly in the immediate time following the operation, it is estimated that 75% of patients experience moderate pain post laparoscopic bariatric surgeries .

Postoperative pain is divided into four types according to cause, Nociceptive Pain is the signal of tissue irritation, impending injury, or actual injury. Neuropathic Pain is the result of the nervous system injury or malfunction, either in the peripheral or in the central nervous system, Psychogenic Pain due to the psychological factors leading to an exaggerated or histrionic presentation of the pain problem, Mixed Category Pain is caused by a complex mixture of nociceptive and neuropathic factors .

Due to the higher risk of respiratory depression, administering opioids to morbidly obese individuals might provide significant challenges when it comes to delivering pain relief .

Acetaminophen is widely considered the cornerstone of perioperative analgesia in the general surgical population.it has been supported by studies and experience in bariatric centers .

Non-steroidal anti-inflammatory drugs (NSAIDs) are components of foundational analgesia for nociceptive pain, which contribute to additional excellent opioid-sparing analgesia. The well-known perioperative concerns with NSAIDs (nephrotoxicity, gastrointestinal (GI) ulceration, and increased bleeding risk) are less likely with cyclooxygenase-2 (COX-2) inhibitors .

Perioperative tramadol side effects in the bariatric surgical population include increased postoperative nausea and vomiting (PONV), serotonin syndrome-inducing interactions (with anti-depressants), and more non-specific intolerance. Despite these, tramadol has been found useful in postoperative pain management after bariatric surgery.

The erector spinae plane block (ESPB) is a kind of paraspinal fascial plane block, which was initially described by Forero et al., (2016). The administration of local anesthetic (LA) occurs in the space between the thoracic transverse processes and the erector spinae muscle. This technique blocks the dorsal and ventral rami of the thoracic and abdominal spinal nerves, resulting in both somatic and visceral sensory blockade. This can potentially provide effective pain relief after abdominal surgery.

ESPB is effective, easy to perform, and can be performed in short time.(13) BUT there is no clear consensus in the studies conducted to determine the optimal level that can be achieved with volume expansion.

Previous reports have mentioned the analgesic effectiveness of one level ESPB in bariatric surgery, but this is the first randomized clinical trial to evaluate the feasibility, efficacy, and safety of two-level bilateral Erector Spinae Plane Block compared to one level in bariatric surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ranges 18 to 60 years old
* Obese patients ; Body mass index(BMI) ≥ 35 - 50 kg/m2
* American Society of Anesthesiologists (13) physical status classes II to III
* Patients scheduled for laparoscopic bariatric surgery i.e. sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB) surgeries

Exclusion Criteria:

* • Refusal of regional block

  * Patients with neurological, psychological disorders or those lacking cooperation.
  * Patients scheduled for concomitant laparoscopic cholecystectomy or paraumbilical hernia repair or those with history of previous bariatric surgery or obstructive sleep apnea.
  * Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
  * Patients with bleeding disorders defined as (INR >1.4) and/ or (platelet count <100,000/µL)
  * Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
  * Patients who are allergic to amide local anesthetics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: included Patient age will range 18 to 60 years, Body mass index(BMI) ≥ 35 - 50 kg/m2, American Society of Anesthesiologists physical status classes II to III, scheduled for laparoscopic bariatric surgery i.e. sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB) surgeries, with normal coagulation profile, npt allergic to amide
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
• Comparison of mean visual analog scale scores at 24 hours postoperative between study groups | 24 hours

SECONDARY OUTCOMES:
Time for first rescue analgesia in both groups | 24 hours
b) Total opioid consumption in both groups in 24hr postoperative | 24 hours
Failure rate in performing the block | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medecine Cairo Uneversity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No